CLINICAL TRIAL: NCT00388310
Title: Effective Duration of Antibiotic Treatment of Community-Acquired Methicillin-Resistant Staphylococcus Aureus (MRSA)
Brief Title: Effective Antibiotic Treatment of MRSA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Christiana Care Health Services (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 26018
Record Dates: First submitted 2006-10-13; First posted 2006-10-16 (Estimated); Last update posted 2012-11-09 (Estimated); Status verified 2012-11

CONDITIONS: Skin Diseases, Infectious
Keywords: cellulitis; furuncles; carbuncles; abscess
MeSH Terms: conditions — Skin Diseases, Infectious; Cellulitis; Furunculosis; Carbuncle; Abscess | interventions — Culture Techniques

ARMS (4):
- Cephalexin (Active Comparator): Cephalexin 250 mg PO q6h x5 days
  Interventions: Procedure: Culture
- Clindamycin (Active Comparator): Clindamycin 300 mg PO q6h x5 days
  Interventions: Procedure: Culture
- trimethoprim/sulfamethoxazole (Active Comparator): trimethoprim/sulfamethoxazole 160 mg/800 mg PO q12h x 5 days
  Interventions: Procedure: Culture
- Placebo (Placebo Comparator)
  Interventions: Procedure: Culture

INTERVENTIONS:
Procedure: Culture — Culture

SUMMARY:
To evaluate the effective duration (in days) to clinical improvement of outpatient antibiotic regimens in the treatment of superficial abscesses caused by MRSA in patients that present to the emergency department.

DETAILED DESCRIPTION:
Skin and soft tissue infections-cellulitis, furuncles, carbuncles, and abscesses-make up approximately 1-2% of emergency room visits annually. While abscesses are generally incised and drained, there is no definite standard treatment regimen or duration of treatment that practitioners have adhered to regarding antibiotic use. Historical evidence suggests that antibiotics may not be necessary for simple superficial abscesses, though a number of antibiotics-including penicillins and cephalosporins-may be used for treatment of large and/or complicated abscesses. These antibiotics however are ineffective against what is becoming an increasingly common pathogen- community-acquired methicillin-resistant Staphylococcus aureus (CA-MRSA).

At our institution, it is estimated that 60-70% (unpublished observation) of cultured abscesses are caused by CA-MRSA. These patients have generally been treated with incision and drainage, with the addition of an antibiotic left to the practitioner's discretion. Also, there has been no universally accepted duration of treatment established to observe clinical improvement of such abscesses. Common antibiotic regimens range from 7-14 days of treatment for cellulitic infections. While there has been one prospective trial regarding the use of antibiotics in simple abscesses, there has been no published prospective study on the use of antibiotics in treating CA-MRSA abscesses in adults. Furthermore, while 7-14 days of treatment seems the recommended duration of treating cellulitic infections, no study has evaluated the duration of treatment needed to observe clinical improvement of abscesses caused by CA-MRSA. We wish to prospectively evaluate the duration of treatment necessary to observe clinical improvement of abscesses caused by CA-MRSA among multiple different antibiotics (ie. cephalexin, clindamycin, and trimethoprim/sulfamethoxazole) after standard incision and drainage in patients presenting to the emergency department.

ELIGIBILITY:
Inclusion Criteria:

* All patients age 18 and older, presenting to the emergency department with an abscess with a diameter greater than three centimeters
* Informed consent

Exclusion Criteria:

* Patients who are presumed to have community-acquired pathogens
* Under 18
* Abscess less than three centimeters in diameter

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2006-02; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
To determine the effective duration of treatment of different antibiotic regimens in the treatment of abscess with regards to resolution of patient symptoms and signs. | 5 days
Treatment failure will be defined as an increase in patient symptoms, increase in abscess size, development of constitutional symptoms, or hospitalization secondary to abscess complications | 5 days

CONTACTS AND LOCATIONS:
Overall Officials: Brian Levine, MD, Principal Investigator — Christiana Care Health Services
Locations (1):
- Christiana Care Health Services, Newark, Delaware, United States